CLINICAL TRIAL: NCT01599988
Title: A Randomised, Double-blinded Study to Compare Milk Protein Isolate (MPI)With Caseinate in Terms of Protein Utilization in Healthy Elderly Subjects
Brief Title: Study to Compare Milk Protein Isolate (MPI) With Caseinate in Terms of Protein Utilization
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Andrea Doolan, Human Studies Manager, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: APC032
Record Dates: First submitted 2012-03-13; First posted 2012-05-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Enteral Feeds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milk protein isolate (Active Comparator): The test meal is a vanilla flavoured enteral drink, containing 1.5kcal/ml, 21% CHO, 6% protein and 5% fat. The 6% protein in this test meal is Milk Protein Isolate.
  Interventions: Dietary Supplement: Milk Protein Isolate
- Caseinate (Active Comparator): The test meal is a vanilla flavoured enteral drink, containing 1.5kcal/ml, 21% CHO, 6% protein and 5% fat. The 6% protein in this test meal is Caseinate.
  Interventions: Dietary Supplement: Caseinate

INTERVENTIONS:
Dietary Supplement: Caseinate — The test meal is a vanilla flavoured enteral drink, containing 1.5kcal/ml, 21% CHO, 6% protein and 5% fat. The 6% protein in this test meal is Caseinate
  Arms: Caseinate
Dietary Supplement: Milk Protein Isolate — The test meal is a vanilla flavoured enteral drink, containing 1.5kcal/ml, 21% CHO, 6% protein and 5% fat. The 6% protein in this test meal is Milk Protein Isolate.
  Arms: Milk protein isolate

SUMMARY:
The Clinical Research Ethics Committee, Cork comprises of faculty representatives, external representatives, legal representatives and appropriate individuals and ex-officio administrative members with needed expertise. Ethics Committee members, including the Chair, are appointed by the Head of College, University College Cork, Medical School.

The Ethics Committee meets once a month.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent.
2. Be between 65 and 75 years of age.
3. Be in generally good health as determined by the investigator.
4. Have no evidence of gastrointestinal disease or of a functional gastrointestinal disorder as determined by the Bowel Disease Questionnaire.
5. Have a stable body weight over the past 3-months.
6. Have a Body Mass Index (BMI) greater than 22, for males and 20 for females and less than 30.
7. Have a satisfactory nutritional status.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 65 and greater than 75 years of age.
2. Have evidence of gastrointestinal disease or other functional gastrointestinal disorder as determined by the Bowel Disease Questionnaire.
3. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic or any condition which contraindicates, in the investigators judgement, entry to the study).
4. Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include anti-inflammatory drugs, corticosteroids, laxatives, enemas, antibiotics (within 1 month), anti-coagulants, and over-the counter non-steroidal analgesics. Subjects should have a wash-out period of two-weeks.
5. Be a smoker.
6. Consume more than the recommended alcohol guidelines i.e. 3-4 alcohol units a day for a man and for a woman 2-3 units a day.
7. Suffer from psychiatric disease
8. Prior gastrointestinal surgery (apart from appendicectomy and hernia repair) or recent unexplained bleeding.
9. Have dietary habits (slimming or vegetarian diet) which could interfere with the assessment of the study product.
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
11. Subjects may not be receiving treatment involving experimental drugs.
12. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
13. Have a malignant disease or any concomitant end-stage organ disease

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Protein utilization | Up to 8 hours

SECONDARY OUTCOMES:
Blood glucose concentrations | Up to 8 hours
Plasma insulin levels | Up to 8 hours
Serum triglycerides | Up to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, MD, BSc, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Ireland